CLINICAL TRIAL: NCT05935176
Title: Phase IV Clinical Trial of Immunogenicity of ACYW135 Meningococcal Polysaccharide Conjugate Vaccine (CRM197 Vector) in a Population Aged 6 to 23 Months
Brief Title: Phase IV Clinical Study of Immunogenicity of ACYW135 Group Meningococcal Polysaccharide Conjugate Vaccine (CRM197 Vector)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CTP-MCVF-004
Record Dates: First submitted 2023-06-27; First posted 2023-07-07 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2024-12

CONDITIONS: Epidemic Meningitis
Keywords: ACYW135; CRM197; Immunogenicity; Persistence; 6~23 months of age
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine Group A (Experimental): 2 dose of ACYW135 group meningococcal polysaccharide conjugate vaccine(MCV4) (0.5ml)
  Interventions: Biological: MCV4
- Vaccine Group B (Experimental): 2 dose of (MCV4) (0.5ml)
  Interventions: Biological: MCV4

INTERVENTIONS:
Biological: MCV4 — 2 dose of MCV4 on Day 0 and Month 1
  Arms: Vaccine Group A
Biological: MCV4 — 2 dose of MCV4 on Day 0 and Month 3
  Arms: Vaccine Group B

SUMMARY:
ACYW135 group meningococcal polysaccharide conjugate vaccine produced by Conchino Biologicals JSC is a covalent coupling conjugate of purified meningococcal podococcal polysaccharide of groups A, C, Y and W135 with CRM197 protein of diphtheria bacillus non-virulent mutant. The purpose of this clinical study is to evaluate the immunogenicity and immunopersistence of the ACYW135 meningococcal polysaccharide conjugate vaccine (CRM197 vector).

DETAILED DESCRIPTION:
Meningococci are divided into 12 serogroups, and 95% of meningococcal cases are caused by serogroups A, B, C, X, W, and Y. Meningococcal epidemic flora can change, and the reasons are related to various factors such as meningococcal strain variation, human mobility transmission, and vaccination against different serogroups of meningococci, etc. The emergence of new serogroups of meningococci can cause the original vaccine to lose its immune protective efficacy and require a new vaccine immunization prevention strategy. the ACYW135 group meningococcal polysaccharide conjugate vaccine was approved in 2016 for a whole population The vaccine has been approved by the State Drug Administration for the prevention of epidemic meningoencephalitis caused by meningococci of groups A, C, W135 and Y in children from 3 months to 3 years of age (47 months of age).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 23 months at the time of screening
* Volunteers who have not received any vaccine containing a epidemic encephalitis component or who have received only the group A polysaccharide flu vaccine and have been vaccinated more than 6 months since their last vaccination. 6 months or more between the last vaccination and the last vaccination
* The legal guardian or delegate has given informed consent, voluntarily signed the informed consent form, and is able to comply with the requirements of the clinical study protocol

Exclusion Criteria:

* Fever before inoculation, axillary temperature >37.0℃
* History of epilepsy, convulsions or seizures or history of psychiatric disorders or family history
* During an acute illness episode; with a serious chronic illness or a condition that is in a progressive stage that cannot be smoothly controlled (or an acute episode)
* Known allergy to a component of the vaccine, especially to diphtheria toxoid
* Live attenuated vaccine received within 14 days or other vaccine received within 7 days prior to enrollment
* Other circumstances that, in the judgment of the investigator, make participation in this clinical study inappropriate
* Those who had a severe allergic reaction after the previous dose of vaccine
* Those with serious adverse reactions causally related to the previous dose of vaccination
* Newly identified or newly occurred cases after the first vaccination that do not meet the inclusion criteria for the first dose or meet the exclusion criteria for the first dose will be determined by the investigator whether to continue to participate in the study

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 660 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Antibody positivity for A, C, Y and W135 in all subjects 6 months after 2 dose exemption | 6 months after 2 dose exemption

SECONDARY OUTCOMES:
Antibody positivity for A, C, Y and W135 in all subjects 9 months after 2 dose exemption | 9 months after 2 dose exemption
A, C, Y and W135 antibody positive conversion rate, positivity rate, GMT, GMI, ≥1:128 ratio in all subjects at 30 days after dose 2 exemption | 30 days after dose 2 exemption
A, C, Y and W135 antibody GMT, GMI, ≥1:128 ratio in all subjects at 6 and 9 months after 2 dose exemption | 6 and 9 months after 2 dose exemption
A, C, Y and W135 antibody GMT, positivity rate, GMI 30 days, 60 days after the first dose, and before the second dose in some subjects of the (0, 3) month immunization program | 30 days , 60 days after the first dose, and before the second dose

CONTACTS AND LOCATIONS:
Locations (1):
- Wuzhi County Center for Disease Control and Prevention, Jiaozuo, Henan, China